CLINICAL TRIAL: NCT05911516
Title: Effects of Pennisetum Purpureum Health Food Supplementation on Muscle Mass and Muscle Strength
Brief Title: Pennisetum Purpureum in Sarcopenia Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202305092
Record Dates: First submitted 2023-05-26; First posted 2023-06-22 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Intervention Model Description: Participants were assigned to either the experimental (n=20) or placebo (n=20) group according to their body composition, upper arm circumference, and lower thigh circumference.
Who Masked: Participant, Investigator
Masking Description: A double-blind, matched-pair study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pennisetum purpureum group (Experimental)
  Interventions: Dietary Supplement: Pennisetum purpureum
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Pennisetum purpureum — 300mg Participants received 900mg of Pennisetum purpureum orally daily for 12 weeks
  Arms: Pennisetum purpureum group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The purpose of this study was to investigate the effects of Pennisetum purpureum health food supplementation on muscle mass and muscle strength.

DETAILED DESCRIPTION:
All participants performed anthropometric measurements (body height, body weight, BMI, blood pressure, body composition, upper arm circumference, and lower thigh circumference), blood collection (hormones, liver function, and kidney function), exercise test (grip strength and 10-m walking test), as well as questionnaire survey before supplementation. Participants were assigned to either the experimental (n=20) or placebo (n=20) group according to their body composition, upper arm circumference, and lower thigh circumference. The definition of insufficient muscle mass was based on the Asian working group for sarcopenia (AWGS) that skeletal muscle mass in extremities by dual-energy X-ray absorptiometry less than 7.0 kg/m2 in men and less than 5.4 kg/m2 in women is a necessary condition, and one of the following criteria were met: (1) handgrip strength less than 28 kg in men and less than 18 kg in women and (2) 5-time chair stand test over than12 seconds. The anthropometric measurements (body height, body weight, BMI, blood pressure, body composition, upper arm circumference, and lower thigh circumference), blood collection (hormones, liver function, and kidney function), exercise test (grip strength and 10-m walking test), as well as questionnaire survey, were collected after 8 weeks and 12 weeks of supplementation.

ELIGIBILITY:
Inclusion Criteria:

1. adult between 18-75 years old
2. skeletal muscle mass in extremities by dual-energy X-ray absorptiometry less than 7.0 kg/m2 in men and less than 5.4 kg/m2 in women
3. one of the following criteria were met: (1) handgrip strength less than 28 kg in men and less than 18 kg in women and (2) 5-time chair stand test over than 12 seconds

Exclusion Criteria:

1. The volunteers have history of cardiovascular, liver, kidney, and diabetes mellitus
2. acute sport injury
3. participated in any clinical trials or experimental research in the last 3 months before our experiment
4. taking supplement during the experimental period
5. did not maintain their regular eating habit or drink alcohol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Body height | Baseline (before supplementation)
Body height | 8 weeks of supplementation
Body height | 12 weeks of supplementation
Body weight | Baseline (before supplementation)
Body weight | 8 weeks of supplementation
Body weight | 12 weeks of supplementation
BMI (body mass index) | Baseline (before supplementation)
BMI (body mass index) | 8 weeks of supplementation
BMI (body mass index) | 12 weeks of supplementation
Systolic blood pressure | Baseline (before supplementation)
Systolic blood pressure | 8 weeks of supplementation
Systolic blood pressure | 12 weeks of supplementation
Diastolic blood pressure | Baseline (before supplementation)
Diastolic blood pressure | 8 weeks of supplementation
Diastolic blood pressure | 12 weeks of supplementation
ASM (Appendicular Skeletal Muscle Mass) | 12 weeks of supplementation
ASM (Appendicular Skeletal Muscle Mass) | 8 weeks of supplementation
Upper Arm Circumference | Baseline (before supplementation)
Upper Arm Circumference | 8 weeks of supplementation
Upper Arm Circumference | 12 weeks of supplementation
Thigh Circumference | Baseline (before supplementation)
Thigh Circumference | 8 weeks of supplementation
Thigh Circumference | 12 weeks of supplementation
Grip Strength | Baseline (before supplementation)
Grip Strength | 8 weeks of supplementation
Grip Strength | 12 weeks of supplementation
10-Meter Walk Test | Baseline (before supplementation)
10-Meter Walk Test | 8 weeks of supplementation
10-Meter Walk Test | 12 weeks of supplementation
Testosterone level | Baseline (before supplementation)
Testosterone level | 8 weeks of supplementation
Testosterone level | 12 weeks of supplementation
Cortisol level | Baseline (before supplementation)
Cortisol level | 8 weeks of supplementation
Cortisol level | 12 weeks of supplementation
Growth Hormone level | Baseline (before supplementation)
Growth Hormone level | 8 weeks of supplementation
Growth Hormone level | 12 weeks of supplementation
Insulin-like Growth Factor-1 | Baseline (before supplementation)
Insulin-like Growth Factor-1 | 8 weeks of supplementation
Insulin-like Growth Factor-1 | 12 weeks of supplementation
follistain level | Baseline (before supplementation)
follistain level | 8 weeks of supplementation
follistain level | 12 weeks of supplementation
myostain level | Baseline (before supplementation)
myostain level | 8 weeks of supplementation
myostain level | 12 weeks of supplementation

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan